CLINICAL TRIAL: NCT01740141
Title: Plexus Brachialis Block. Better to do by Start Than by End of Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Holmberg, Principal investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/476a
Record Dates: First submitted 2012-11-22; First posted 2012-12-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plexus before surgery (Other): Plexus brachialis before surgery
  Interventions: Procedure: Plexus brachialis block
- Plexus after surgery (Other): Plexus brachialis performed after surgery
  Interventions: Procedure: Plexus brachialis block

INTERVENTIONS:
Procedure: Plexus brachialis block
  Other Names: LSIB. Ropivacain 7,5 mg/ml, 0,5 ml/kg

SUMMARY:
The aim of the study is to find out if the timing of brachial plexus block, before or after surgery, has an impact of the extent of acute postoperative surgical pain or the incidence and severity of long-lasting (chronic) pain after surgery.

This is a prospective, randomized, double blind study in patients with radial fractures undergoing surgery with volar plate. The patients will be followed up for 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Radial fracture
* ASA 1 and 2
* Able to communicate in norwegian
* Suitable for surgery in general anaesthesia and brachial plexus block

Exclusion Criteria:

* Pregnancy
* Chronic pain
* BMI over 35

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain | postoperative to 6 months
  NAS

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holmberg, MD, Principal Investigator — MD Ullevaal sykehus
Locations (1):
- Oslo Universitetssykehus, Ullevaal, dept of anaesthesiology, legevakten, Oslo, Oslo County, Norway